CLINICAL TRIAL: NCT06838143
Title: Real Life Non-interventional Study on Safety and Effectiveness of Ilaris® (Canakinumab) 150 mg for Subcutaneous Injection in Hereditary Periodic Fever Syndrome (CAPS, crFMF, TRAPS and HIDS/MKD) Patients and sJIA Patients (REASSURE)
Brief Title: Ilaris NIS in Korea
Acronym: REASSURE
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CACZ885NKR01
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Periodic Fever Syndromes; Cryopyrin-associated Periodic Syndromes (CAPS); Colchicine Resistance Familial Mediterranean Fever (crFMF); TNF Receptor Associated Periodic Syndrome (TRAPS); Hyper-IgD Syndrome / Mevalonate Kinase Deficiency (HIDS/MKD); Systemic Juvenile Idiopathic Arthritis (sJIA)
Keywords: Hereditary Periodic Fever Syndromes; Cryopyrin-associated periodic syndromes (CAPS); colchicine resistance familial Mediterranean fever (crFMF); TNF receptor associated periodic syndrome (TRAPS); Hyper-IgD syndrome / Mevalonate kinase deficiency (HIDS/MKD); Systemic juvenile idiopathic arthritis (sJIA)
MeSH Terms: conditions — Hereditary Autoinflammatory Diseases; Cryopyrin-Associated Periodic Syndromes; Periodic fever, familial, autosomal dominant; Mevalonate Kinase Deficiency; Arthritis, Juvenile | interventions — canakinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Ilaris: Patients treated with Ilaris in a clinical setting
  Interventions: Biological: Ilaris

INTERVENTIONS:
Biological: Ilaris — Prospective observational study. There is no treatment allocation.

SUMMARY:
This is a study to evaluate safety and effectiveness of Ilaris in adult and pediatric patients receiving the drug in a clinical setting for any of the following indications, Hereditary Periodic Fever Syndromes, Cryopyrin-associated periodic syndromes (CAPS), colchicine resistance familial Mediterranean fever (crFMF), TNF receptor associated periodic syndrome (TRAPS), Hyper-IgD syndrome / Mevalonate kinase deficiency (HIDS/MKD) or Systemic juvenile idiopathic arthritis (sJIA).

DETAILED DESCRIPTION:
This is a prospective observational, multicenter, uncontrolled, open-label non-interventional study in ≥2 year and <19 year-old pediatric and ≥19 year-old adult hereditary periodic fever syndrome patients and ≥2 year and <19 year-old sJIA patients receiving Ilaris for the treatment of CAPS, crFMF, TRAPS, HIDS/MKD and sJIA, respectively, partially using retrospective observation to collect and evaluate data on the safety and effectiveness of Ilaris in patients receiving this drug in a clinical setting for any of these indications. The whole study period is up to 4 years, consisting of a 2-year enrollment period and 2-year observation period.

As all pediatric and adult hereditary periodic fever syndrome patients and all sJIA patients receiving Ilaris for approved indications will be enrolled, this study has no fixed sample size.

For subjects who started Ilaris before enrolling in this study, the safety and effectiveness baseline and early period data will be retrospectively collected.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent/assent of the patient or their legal representative/parent (≥2 year and <19 year-old pediatric patient) for voluntarily participating in this study
2. Age: ≥2 year and <19 year-old pediatric and ≥19 year-old adult hereditary periodic fever syndrome (CAPS, crFMF, TRAPS and HIDS/MKD) patients and ≥2 year and <19 year-old sJIA patients
3. Patient who have an agreement to be treated or who have already started treatment with Ilaris in accordance with the approved label information

Exclusion Criteria:

1. Patients receiving Ilaris treatment for autoimmune disease other than CAPS, crFMF, TRAPS, HIDS/MKD or sJIA
2. Patients participating in an interventional clinical trial which would have an impact on routine clinical treatment

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ≥2 year and <19 year-old pediatric and ≥19 year-old adult hereditary periodic fever syndrome patients and ≥2 year and <19 year-old sJIA patients receiving Ilaris for the treatment of CAPS, crFMF, TRAPS, HIDS/MKD and sJIA
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-03-29 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | Up to 104 weeks from Ilaris treatment
  Adverse events and serious adverse events in hereditary periodic fever syndrome (CAPS, crFMF, TRAPS and HIDS/MKD) and sJIA patients treated with Ilaris.

SECONDARY OUTCOMES:
Proportion of complete responders | Up to 16 weeks from Liars treatment
  Defining patients as responders when they are assessed as having achieved complete response at 4 weeks of treatment and reach 16 weeks of treatment without flare for crFMF, TRAPS, HIDS/MKD and sJIA patients or complete response at 8 weeks of treatment and reach 16 weeks of treatment without flare for CAPS patients.
  Complete response will be evaluated in patients with data of clinical response as measured by Physician Global Assessment of Disease Activity (PGA) (5-point scale of none, minor, mild, moderate and severe) Complete response is defined as meeting both of the following criteria.
  * PGA ≤ minor (PGA < 2) (clinical response)
  * CRP ≤10 mg/L (= 1 mg/dL), or reduction by ≥70% from the start of treatment (serological response) Flare is defined as meeting both of the following criteria.
  * PGA ≥ mild (PGA ≥ 2) (clinical flare)
  * CRP >30 mg/L (= 3 mg/dL) (serological flare)
Proportion of participants with Physician Global Assessment of Disease Activity (PGA) score <2 | Up to 104 weeks from Ilaris treatment
  Participants assessed by physician on Physician's Global Assessment measured on a 5--point scale for disease activity as: 0 = None/absent; 1 = Minor; 2 = Mild; 3 = Moderate; 4 = Severe.
Proportion of patients with C- reactive protein (CRP) serological response | Up to 104 weeks from Ilaris treatment
  Proportion of patients with a C-reactive protein (CRP) of ≤ 10 mg/L or a ≥ 70% decrease from the start of treatment.
Proportions of patients with serum amyloid A (SAA) normalization | Up to 104 weeks from Ilaris treatment
  Proportions of patients with serum amyloid A (SAA) normalization defined as SAA ≤ 10 mg/L.
Proportion of patients classified in each severity level in the physician's severity assessment of key disease -specific signs and symptoms | Up to 104 weeks from Ilaris treatment
  Physician's severity assessment of key disease-specific signs/symptoms uses the following 5- point scale.
  0 = none
  1. = minor
  2. = mild
  3. = moderate
  4. = severe Key signs/symptoms to be assessed differ from disease to disease under study, which are as follows.
  CAPS: hearing impairment, visual impairment, renal impairment, and joint dysfunction, skin rash, injection site reaction crFMF: chest pain, abdominal pain, arthralgia/arthritis, skin rash TRAPS: skin rash, musculoskeletal pain, abdominal pain, eye manifestations HIDS (MKD): lymphadenopathy, aphthous ulcers, abdominal pain sJIA: arthritis, generalized lymphadenopathy, rheumatoid rash, hepatosplenomegaly or splenomegaly, serositis
Proportions of patients classified in each severity level in symptoms likely to significantly affect affect physical functioning and vital prognosis | Up to 104 weeks from Ilaris treatment
  Symptoms that may significantly affect physical functioning and vital prognosis will be evaluated using the following 5-point scale.
  0 = none
  1. = minor
  2. = mild
  3. = moderate
  4. = severe Evaluation of auditory disorder, visual disorder and renal impairment, and status of central nervous system disorder
Percent change from baseline in Health related quality of life (HRQOL) measured by Child Health Questionnaire-Parent Form 50 (CHQ-PF50) | Up to 104 weeks from Ilaris treatment
  The CHQ is a generic self-administered instrument designed to capture the physical, emotional, and social components of health status of children. It comprises 15 health concepts (range, 0 to 100) exploring either physical and psychosocial domains. Higher scores in the scales indicate better HRQoL.
Percent change from baseline in Health related quality of life (HRQOL) measured by 36-item Short Form Health Survey (SF-36) | Up to 104 weeks from Ilaris treatment
  The SF-36 health survey is a subjective measure of health-related QoL and consists of 36 questions relating to eight domains: physical functioning, social functioning, physical role functioning, emotional role functioning, vitality, mental health, pain, and general health. Scores of each domain varies from 0 to 100 points, and a higher score represents better QoL
Percent change from baseline in Health related quality of life (HRQOL) measured by Work Productivity and Activity Impairment Specific Health Problem v2.0 (WPAI-SHP) | Up to 104 weeks from Ilaris treatment
  The WPAI-SHP contains six items relating to health problems interfering with work or daily activities over the previous week, the WPASI-SHP yields four scores, absenteeism, presenteeism, work productivity loss, and activity impairment, which can range from 0 (no impact on work/activities) to 100 (total incapacity).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No